CLINICAL TRIAL: NCT03277183
Title: Frequent, Low-Dose Erythropoietin: A Mechanistic Approach to Mitigate Adverse Cardiovascular Effects of Erythropoietin Therapy in Patients With Chronic Kidney Disease
Brief Title: Frequent, Low-Dose Erythropoietin A Mechanistic Approach to Mitigate Adverse Cardiovascular Effects of Erythropoietin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CARA-019-16F; I01CX001449 (NIH)
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Anemia; CKD; Atherosclerosis; Cardiovascular
Keywords: erythropoietin
MeSH Terms: conditions — Anemia; Atherosclerosis | interventions — Erythropoietin; Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned two different erythropoietin dosing strategies. One group will be given more frequent, low-doses of EPO and the other group will be given the same, cumulative dose given every 2 weeks.
Who Masked: Outcomes Assessor
Masking Description: The outcome is the progression of carotid plaque. John Forder, PhD, who will read the MRIs will be blinded to the subject and treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low dose erythropoietin (Placebo Comparator): Subjects randomized to this arm will receive low-dose of EPO administered thrice weekly
  Interventions: Drug: Low dose erythropoietin
- High dose erythropoietin (Experimental): Subjects randomized to this arm will receive the same cumulative dose of EPO administered as a high-dose of EPO every 2 weeks
  Interventions: Drug: High dose erythropoietin

INTERVENTIONS:
Drug: Low dose erythropoietin — Subjects randomized to this arm will receive low-dose of EPO administered thrice weekly
  Other Names: Low dose
  Arms: Low dose erythropoietin
Drug: High dose erythropoietin — Subjects randomized to this arm will receive the same cumulative dose of EPO administered as a high-dose of EPO every 2 weeks
  Other Names: High dose
  Arms: High dose erythropoietin

SUMMARY:
Although several large well designed clinical trials have shown that erythropoietin which is commonly used to treat anemia associated with kidney disease, increases the risk of stroke and heart disease, the mechanism for this increased risk is unknown. The investigators' preliminary studies show that the adverse effects of erythropoietin are from activation of the heterodimeric erythropoietin/ beta common receptor which only occurs with high doses of erythropoietin. The investigators propose a clinical trial of 120 patients assigned to low doses of erythropoietin given more frequently or the same cumulative dose of erythropoietin administered as a high dose once every two weeks and assess effects on the beta common receptor activation, inflammation and vascular disease as evidence by MRI of the carotid arteries.

DETAILED DESCRIPTION:
Erythropoietin (EPO) is the most widely prescribed cytokine, yet the benefits and potential side effects of different dosing regimens are poorly understood. It is now recognized that erythropoietin administered at high doses to patients with chronic kidney disease, results in an increased risk of morbidity and mortality from heart disease and stroke. However, the mechanisms that mediate this increased risk of cardiovascular disease is not known. There are two receptors for erythropoietin the homodimeric EPO receptor (EPOR) and the heterodimeric beta common receptor ( CR)/EPOR. The investigators have demonstrated that activation of the heterodimeric CR/EPOR only occurs with high doses of EPO. Our exciting, published, preliminary data also demonstrates that the CR is in a complex with vascular endothelial growth factor receptor-2 (VEGFR-2) and that high doses of EPO activate VEGFR-2 through the CR, resulting in the deleterious effects of VEGFR-2 activation on the cardiovascular system. This is particularly important in patients with kidney disease since they are already at a high risk of cardiovascular disease. Moreover in advanced kidney disease cyanate derived from the high urea levels can non-enzymatically form an amide bond with EPO. This carbamylated EPO (cEPO) has no effect on hemoglobin, but still activates the heterodimeric CR/EPOR. To date there have been no studies that have directly measured levels of cEPO or activation of the CR/EPOR in patients with kidney disease. Our hypothesis is that the administration of low-doses of EPO more frequently will result in lower levels of total and carbamylated erythropoietin decreased activation of VEGFR-2 via the heterodimeric CR/EPOR and consequently decreased inflammation and atherosclerosis. The investigators will directly test this hypothesis by randomly allocating 120 patients with chronic kidney disease to either low- dose EPO given thrice weekly or the same cumulative dose, a high-dose, administered once every 2 weeks. Our hypothesis predicts that low-dose EPO will be as effective at correcting anemia, but will demonstrate less progression of carotid artery plaque, as assessed by non-contrast magnetic resonance imaging, as compared to the high-dose, EPO given every 2 weeks. To delineate how EPO affects blood vessels, the investigators will isolate endothelial cells from blood vessels in 20 patients who are assigned to low-dose EPO and 20 allocated to high-dose EPO. Within these cells the investigators will investigate the signaling pathways that are triggered by activation of CR/EPOR. In a substudy of 20 subjects with kidney disease randomized to low-dose EPO or to high-dose EPO, as well as 20 healthy controls receiving a single dose of high- or low-dose EPO, the investigators will determine how kidney function and dosing affects levels of total and carbamylated erythropoietin. The investigators' study will not only provide us with a thorough understanding of the mechanism by which EPO mediates the increased risk of atherosclerosis, but a clinical strategy to avoid the side effects of EPO therapy and a tool to quantify the cardiovascular risk of EPO and newer erythropoiesis stimulating agents by assessing activation of the heterodimeric CR/EPOR.

ELIGIBILITY:
Inclusion Criteria:

The investigators will enroll Veterans who fulfill the following criteria:

* stage 3, 4, or 5 CKD (estimated glomerular filtration rate of less than 60 ml/min/1.73 m2) on at least two separate occasions greater than 3 months apart; and
* candidates for EPO therapy as per the National Kidney Foundation's Kidney Disease Outcomes Quality Initiative guidelines (hemoglobin < 10 gm/dL and anemia of CKD).

Exclusion Criteria:

The investigators will exclude any Veteran who meets any of the following criteria:

1. pregnant, planning to become pregnant in the next year, or breast feeding;
2. uncontrolled hypertension (blood pressure > 180/100 mm Hg despite optimal antihypertensive medications);
3. active gastrointestinal bleeding (visible blood or positive tests for stool occult blood accompanied by a decrease in hemoglobin);
4. likely to have EPO resistance;
5. an adverse cardiovascular event in the prior three months;
6. active or recent (within the last 3 months) severe, systemic infection;
7. active inflammatory disease such as lupus, rheumatoid arthritis, or vasculitis requiring immunosuppressive or immunomodulatory medications;
8. history of solid organ transplantation;
9. expected off-dialysis survival of less than one year (as determined by the estimated glomerular filtration slope and the treating physician;
10. active cancer (undergoing chemotherapy or radiation within the last 3 months) or primary bone marrow disease such as myelofibrosis; or
11. a contraindication for an MRI or individuals who cannot comply with the study protocol. The investigators will exclude healthy subjects that meet a, b, f, g, h, or j.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Segal, MD PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Erythropoietin | High Dose Erythropoietin
Started | 3 | 2
Completed | 0 | 0
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: Although baseline MRI's were performed they were not analyzed due to study termination due to lack of enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Erythropoietin | High Dose Erythropoietin | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 68 (5) | 67 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Carotid Total Plaque Volume From Baseline to Approximately 1 Year, as Assessed by Non-contrast MRI
Description: The plaque characteristics will be analyzed by MRI-PlaqueViewTM (VP diagnostics Inc., WA). Planimetry will be performed on the image data sets, using histogram equalization to improve edge detection for plaque, arterial wall and lumen. Differences in image contrast between T1-weighted, T2-weighted, Time of Flight, and proton density will be used to characterize the plaque as fibrous, stable, or unstable.
Time Frame: 1 year
Population: Since the study was terminated due to lack of enrollment and the paperwork to obtain the software to read the MRI was still being filled out, we did not have the software to analyze the MRI and thus there is no data to report.
Arm/Group | Low Dose Erythropoietin | High Dose Erythropoietin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Severity of Maximal Stenosis at Baseline and Upon Follow-up.
Description: as for outcome 1
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Low Dose Erythropoietin | High Dose Erythropoietin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Total Plaque Area at Baseline and Upon Follow-up.
Description: as for outcome 1
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Low Dose Erythropoietin | High Dose Erythropoietin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Characteristics of Plaques (Soft or Fibrous and Stable or Unstable) at Baseline and Upon Follow-up.
Description: as for outcome 1
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Low Dose Erythropoietin | High Dose Erythropoietin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The time period of adverse events where for the time that each subject was enrolled in the study. No study completed the study since the study was closed prematurely.
Arm/Group | Low Dose Erythropoietin | High Dose Erythropoietin
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT03277183/Prot_SAP_000.pdf